CLINICAL TRIAL: NCT04746781
Title: The Effect of Mobile Immersive Video and Motivation and Problem Solving on Enrollment in the Diabetes Prevention Program
Brief Title: The Effect of 360 Video and MAPS on Enrollment in the DPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Bryan Smith Gibson, Assistant Professor Biomedical Informatics, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00132307
Record Dates: First submitted 2021-02-01; First posted 2021-02-10 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus, Type 2; PreDiabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Risk notification/education arm (Active Comparator): We will send all participants a short message service (SMS) message with a link to a website that educates the public about their risk for developing T2DM and about the availability and efficacy of the DPP to address their risk
  Interventions: Behavioral: Risk notification/education
- Mobile 360° Video intervention arm (Experimental): After risk notification and education, participants will receive links to two 3-minute immersive Mobile 360° Videos (in which the viewer moves their phone to 'look around' the world of the video) on their smart phones. These videos are intended to influence affective and experiential perceptions of risk. The first video tells an emotional story of the negative effects on an individual's health and family life as they progress from prediabetes to T2DM and develop cardiovascular complications. The second video provides the viewer with a vicarious experience of the changes in vision that occur as diabetic retinopathy develops and worsens.
  Interventions: Behavioral: Mobile 360° Video intervention; Behavioral: Risk notification/education
- Motivation and Problem Solving (MAPS) arm (Experimental): After risk notification and education, participants will be called by a health coach trained in counseling/coaching. The coach will guide them in setting goals related to their health, and addressing any practical barriers to enrolling/engaging in the DPP if that is consistent with their health goals. Per their preference, participants will receive up to 5 phone calls from the health coach over a 4 week period.
  Interventions: Behavioral: Motivation and Problem Solving (MAPS); Behavioral: Risk notification/education

INTERVENTIONS:
Behavioral: Mobile 360° Video intervention — Using 360° Videos to educate participants about the effect of diabetes.
  Arms: Mobile 360° Video intervention arm
Behavioral: Motivation and Problem Solving (MAPS) — Using Motivation and Problem Solving to help people enroll in the Diabetes Prevention Program.
  Arms: Motivation and Problem Solving (MAPS) arm
Behavioral: Risk notification/education — Sending participants (all of whom meet the diagnostic criteria for prediabetes) educational information about the condition.

SUMMARY:
We will conduct a three-armed randomized, clinical trial to test the incremental effectiveness of Mobile 360° Video and Motivation and Problem Solving in motivating individuals with Prediabetes to enroll in the Diabetes Prevention Program. all participants will receive notification that they have Prediabetes and education about Prediabetes, Type 2 diabetes, and the Diabetes Prevention Program, some participants will receive the additional interventions

DETAILED DESCRIPTION:
More than 88 million Americans are at risk of developing Type 2 diabetes mellitus (T2DM). The one-year Diabetes Prevention Program (DPP) has been shown to be effective in reducing the risk of progressing from prediabetes to T2DM. However, most individuals who could benefit from the program never enroll.

Prior research has elucidated several reasons people do not enroll in the DPP. First, many people are not aware that they are at risk of developing T2DM, or that an efficacious program like the DPP exists. Second, the complications from T2DM are abstract, distal and difficult to imagine, which in turn leads to low motivation for risk-reducing behaviors. Finally, practical barriers limit DPP enrollment including cost, travel time, and scheduling. Prior research has tested rational appeals (such as provider-based education and referral) to enroll individuals in the DPP, with limited efficacy. In this project we will compare the effects of notification and education alone, notification and education plus mobile phone delivered videos (emotional appeal), and notification and education plus phone-based coaching utilizing a motivation and problem-solving approach. Our primary outcome will be enrollment and 1-month engagement in the DPP.

This three-armed randomized, clinical trial will be conducted within 2 health systems. Following an opt-out procedure offered to all eligible participants, participants will complete informed consent and a baseline survey. In the risk notification/education arm, we will send all participants a short message service (SMS) message with a link to a website that educates the public about their risk for developing T2DM and about the availability and efficacy of the DPP to address their risk. In the Mobile 360° Video intervention arm, after risk notification/education, participants will receive links to two 3-minute immersive Mobile 360° Videos (in which the viewer moves their phone to 'look around' the world of the video) on their smart phones. These videos are intended to influence affective and experiential perceptions of risk. The first video tells an emotional story of the negative effects on an individual's health and family life as they progress from prediabetes to T2DM and develop cardiovascular complications. The second video provides the viewer with a vicarious experience of the changes in vision that occur as diabetic retinopathy develops and worsens.

In the Motivation and Problem Solving (MAPS) arm, after risk notification/education, participants will be called by a health coach trained in counseling/coaching. The coach will guide them in setting health related goals and addressing any practical barriers to enrolling/engaging in the DPP, if that is consistent with their health goals.

ELIGIBILITY:
Inclusion Criteria:

* Are aged 18-89
* Have a diagnosis of prediabetes within the past 5 years (ICD-10 code R73.03)
* Have an email and mobile telephone number on record with the Health-system
* Primary language of either English or Spanish

Exclusion Criteria:

* Type 2 diabetes mellitus (ICD-10-CM E11);
* Type 1 diabetes mellitus (ICD-10-CM Diagnosis E10),
* Diabetes mellitus due to underlying condition (ICD-10 E08);
* Drug or chemical induced diabetes mellitus (ICD-10 E09);
* Gestational diabetes (ICD-10 024.4);
* Neonatal diabetes mellitus (ICD-10 P70.2);
* Post-pancreatectomy diabetes mellitus (ICD-10 E13).
* Patients whose primary language is other than Spanish or English will be excluded.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 818 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Diabetes prevention program enrollment | 1-month
  Enrollment in the Diabetes prevention program . This data that is recorded by all Diabetes prevention programs and is required to be reported to the Centers for disease control. For individuals attending an in person-class. It is defined by the CDC as registration for the program. For individuals who enroll in an online DPP it is defined by the CDC as an individual setting their password for the app. For the purposes of this trial any individual meeting either of these criteria will be considered to have enrolled in the DPP.
4 weeks of engagement in the Diabetes prevention program | 1 month
  1-month engagement in the Diabetes prevention program. This is data that is recorded by all Diabetes prevention programs and is required to be reported to the Centers for Disease Control. For individuals attending an in person-class, it is defined by the CDC as the individual attending at least 2 of the first four sessions. For individuals who enroll in an online DPP it is defined by the CDC as completing at least two of the following activities: (A) Complete two education modules (B) Send at least 1 In-App message and/or Group Wall post (C) Set or log at least one behavior (D) Log, plan or research at least three meals (E) Log physical activity at least three (F) Weigh-in on three or more days in two out of the first four weeks
  For the purposes of this trial any individual meeting either of these criteria will be considered to have engaged in the DPP for the first month.

SECONDARY OUTCOMES:
Changes in self-efficacy | 1 month
  Self-efficacy related to Diabetes prevention program participation as well as diet, exercise, and weight loss will be measured using the brief (16 items) Self-Efficacy scales adapted from Wilson 2016:
  Wilson KE, Harden SM, Almeida FA, et al. Brief self-efficacy scales for use in weight-loss trials: Preliminary evidence of validity. Psychological assessment 2016; 28(10): 1255-64.
  This will be measured pre and post intervention and the change score calculated and compared across intervention arms
Changes in Risk perceptions | 1 month
  Risk perceptions related to development of Type 2 Diabetes will be measured using an 18-item measure of risk perceptions for Type 2 diabetes developed by Ferrer et al:
  Ferrer RA, Klein WMP, Persoskie A, Avishai-Yitshak A, Sheeran P. The Tripartite Model of Risk Perception (TRIRISK): Distinguishing Deliberative, Affective, and Experiential Components of Perceived Risk. Annals of Behavioral Medicine 2016; 50(5): 653-63.
  This measure includes 6 items each to measure three different aspects of risk perception: deliberative, affective and experiential risk perceptions. we will calculate the sub scores for these dimensions and compare changes in them across intervention arms

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kent-Marvick J, Knysheva M, Gibson B, Simonsen SE. Why Do People Choose to Enroll or Not Enroll in the National Diabetes Prevention Program Lifestyle Change Program? A Mixed-Methods Analysis From a Sample of Adults With a Prediabetes Diagnosis. J Prim Care Community Health. 2024 Jan-Dec;15:21501319241282862. doi: 10.1177/21501319241282862. PMID 39305089
- [Derived] Gibson B, Simonsen S, Barton J, Zhang Y, Altizer R, Lundberg K, Wetter DW. Motivation and Problem Solving Versus Mobile 360 degrees Videos to Promote Enrollment in the National Diabetes Prevention Program's Lifestyle Change Program Among People With Prediabetes: Protocol for a Randomized Trial. JMIR Res Protoc. 2021 Jun 14;10(6):e28884. doi: 10.2196/28884. PMID 34125075